CLINICAL TRIAL: NCT00445718
Title: Perinatal Neuroblastoma: Expectant Observation A Children's Oncology Group Pilot Study
Brief Title: Natural History Study of Infants With Adrenal Masses Found on Prenatal and/or Neonatal Imaging
Status: Completed | Type: Observational
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: ANBL00P2; NCI-2009-00398 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); COG-ANBL00P2 (Other: Children's Oncology Group); U10CA098543 (NIH)
Record Dates: First submitted 2007-03-07; First posted 2007-03-09 (Estimated); Last update posted 2017-02-09 (Estimated); Status verified 2017-02

CONDITIONS: Adrenocortical Carcinoma; Localized Resectable Neuroblastoma; Precancerous Condition
MeSH Terms: conditions — Adrenocortical Carcinoma; Precancerous Conditions

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, Tumor tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observational: Patients undergo an abdominal CT or MRI scan on weeks 0, 6, and 42 and an abdominal sonogram on weeks 0, 3, 6, 12, 18, 30, 42, 66, and 90. Urinary catecholamine levels are also measured on the same weeks as the abdominal sonogram. Patients with an increase in tumor volume or catecholamine levels undergo sonographic evaluation and urine catecholamine sampling every 3 weeks until stabilization. Patients with a continued increase in catecholamine levels or a 50% increase in tumor volume undergo surgical resection off protocol therapy.
  Interventions: Procedure: computed tomography; Procedure: 3-Tesla magnetic resonance imaging; Procedure: Abdominal Sonogram

INTERVENTIONS:
Procedure: computed tomography
  Other Names: tomography, computed
Procedure: 3-Tesla magnetic resonance imaging
  Other Names: 3-Tesla MRI; 3T MRI
Procedure: Abdominal Sonogram — Sonogram of the abdomen area

SUMMARY:
This natural history study is collecting health information about infants with adrenal masses found on prenatal and/or neonatal imaging. Gathering information over time from imaging and laboratory tests of infants with adrenal masses may help doctors learn more about the disease and plan the best treatment.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Determine whether nonoperative management of infants with adrenal masses found on prenatal and/or neonatal imaging results in a 3-year survival rate of 95%.

SECONDARY OBJECTIVES:

I. Estimate the percentage of these patients who are spared surgical resection. II. Evaluate the natural history and histology of perinatal adrenal masses. III. Evaluate the tumor biology and histology of prenatal and neonatal neuroblastomas.

IV. Determine the tumor characteristics that are associated with a need for resection.

OUTLINE:

Patients undergo an abdominal CT or MRI scan on weeks 0, 6, and 42 and an abdominal sonogram on weeks 0, 3, 6, 12, 18, 30, 42, 66, and 90. Urinary catecholamine levels are also measured on the same weeks as the abdominal sonogram. Patients with an increase in tumor volume or catecholamine levels undergo sonographic evaluation and urine catecholamine sampling every 3 weeks until stabilization. Patients with a continued increase in catecholamine levels or a 50% increase in tumor volume undergo surgical resection off protocol therapy.

After a patient goes off-observation, they will be monitored every six months for two years, and annually thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Sonographically identified adrenal mass meeting one of the following criteria:

  * No greater than 16 mL in volume, if solid
  * No greater than 65 mL if at least 25% cystic and does not cross the midline
* Disease limited to the adrenal gland

  * No evidence of positive contralateral or ipsilateral lymph nodes or other spread outside the adrenal gland by CT scan or MRI
  * No evidence of disease outside the adrenal gland by MIBG scan
  * Negative for tumor cells by bone marrow biopsy, if performed
* No more than 6 months of age on the date the mass is first identified
* No prior chemotherapy
* No prior abdominal surgery

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients with sonographically identified adrenal mass
Sampling Method: Non-Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2001-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Survival rate | Up to 3 years
  Estimated using the Kaplan-Meier method.
Event-free survival (EFS) | Up to 3 years
  Estimated using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Jed Nuchtern, MD, Principal Investigator — Children's Oncology Group
Locations (45):
- United States (38):
  - University of Arizona Health Sciences Center, Tucson, Arizona
  - Southern California Permanente Medical Group, Downey, California
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Alfred I duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Baptist Hospital of Miami, Miami, Florida
  - Childrens Memorial Hospital, Chicago, Illinois
  - Advocate Lutheran General Hospital, Park Ridge, Illinois
  - Southern Illinois University, Springfield, Illinois
  - Maine Children's Cancer Program, Scarborough, Maine
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Saint Joseph's Regional Medical Center, Paterson, New Jersey
  - Brooklyn Hospital Center, Brooklyn, New York
  - The Steven and Alexandra Cohen Children's Medical Center of New York, New Hyde Park, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester, Rochester, New York
  - Mission Hospitals Inc, Asheville, North Carolina
  - Children's Hospital Medical Center of Akron, Akron, Ohio
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Rainbow Babies and Childrens Hospital, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - T C Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Childrens Hospital, Knoxville, Tennessee
  - St. Jude Children's Research Hospital, Memphis, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Medical City Dallas Hospital, Dallas, Texas
  - Cook Children's Medical Center, Fort Worth, Texas
  - Baylor College of Medicine, Houston, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Naval Medical Center - Portsmouth, Portsmouth, Virginia
  - Seattle Children's Hospital, Seattle, Washington
  - Providence Sacred Heart Medical Center and Children's Hospital, Spokane, Washington
  - Saint Vincent Hospital, Green Bay, Wisconsin
- Royal Children's Hospital, Parkville, Victoria, Australia
- Canada (6):
  - IWK Health Centre, Halifax, Nova Scotia
  - Chedoke-McMaster Hospitals, Hamilton, Ontario
  - Hospital for Sick Children, Toronto, Ontario
  - Hospital Sainte-Justine, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Ste-Foy, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan

REFERENCES:
- [Derived] Nuchtern JG, London WB, Barnewolt CE, Naranjo A, McGrady PW, Geiger JD, Diller L, Schmidt ML, Maris JM, Cohn SL, Shamberger RC. A prospective study of expectant observation as primary therapy for neuroblastoma in young infants: a Children's Oncology Group study. Ann Surg. 2012 Oct;256(4):573-80. doi: 10.1097/SLA.0b013e31826cbbbd. PMID 22964741